CLINICAL TRIAL: NCT00899366
Title: Molecular Mechanisms of NOTCH Induced Transformation in T-ALL
Brief Title: DNA Analysis of Tissue From Patients With T-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000529758; ECOG-E2993T2 (Other: ECOG-ACRIN); R01CA129382 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: T-cell adult acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Microarray Analysis; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow and blood nucleic acids and cells.

INTERVENTIONS:
Genetic: microarray analysis
Genetic: mutation analysis
Other: immunologic technique

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at tissue samples from patients with T-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify the transcriptional signatures associated with the presence of NOTCH1 mutations in primary T-cell acute lymphoblastic leukemia (T-ALL) cells using oligonucleotide microarrays.
* Characterize the global changes on gene expression resulting from the inactivation of NOTCH signaling in human T-ALL lymphoblasts.

OUTLINE: This is a multicenter study.

Frozen lymphoblast samples from patients with T-cell acute lymphoblastic leukemia (NOTCH1-mutated and wild type) are assessed for genetic expression profiles and mutations by microarray analysis and activated NOTCH1 protein by western blot analysis.

PROJECTED ACCRUAL: A total of 48 samples from patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of T-cell acute lymphoblastic leukemia
* Frozen lymphoblast samples available

  * NOTCH1-mutated or wild type sample available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E2993
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2006-12-28 (Actual); Primary Completion 2009-07-30 (Actual); Study Completion 2009-07-30 (Actual)

PRIMARY OUTCOMES:
Transcriptional signatures associated with NOTCH1 mutations in T-cell acute lymphoblastic leukemia (T-ALL) cells | 1 month
  Mutational analysis
Global changes on gene expression resulting from inactivation of NOTCH signaling in T-ALL cells | 1 month
  Gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo A. Ferrando, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center

REFERENCES:
- See also: Manuscript — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2721784/